CLINICAL TRIAL: NCT00666315
Title: Harmonic FOCUS Versus Conventional Technique in Total Thyroidectomy for Benign Thyroid Disease -A Prospective, Comparative, Multicenter, Observational Study
Brief Title: Harmonic FOCUS Versus Conventional Technique in Total Thyroidectomy for Benign Thyroid Disease
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Prof. Dr. Miccoli, University of Pisa
Other Study IDs: CME-07-001; EO-0469
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Benign Thyroid Disease
Keywords: Consecutive euthyroid patients with multinodular goiter for whom a total Thyroidectomy under general anesthesia is indicated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Harmonic: Group operated with Harmonic device
- Conventional: Group operated with Electrocauery and Clip/Suture

SUMMARY:
New haemostatic techniques have been developed with the advent of laparoscopic surgery. Among other things, ultrasound instruments have been used for the dissection, division and coagulation of vessels and other tissue. Previous studies in Thyroidectomy observed a clinically and economically significant reduction in operating time with no increase in the complication rate when the Harmonic device has been used. The aim of the present clinical trial is to evaluate potential advantages of a new Harmonic device (FOCUS), developed especially for Thyroid procedures, in the use of HS in thyroidectomies when compared with EC in terms of operative time, number of ligatures, QoL, blood loss, pain intensity at the surgical site, amount of drainage, and complications, including the incidence of RLN palsy and hypoparathyroidism.

DETAILED DESCRIPTION:
Thyroidectomy is one of the most frequently performed operations in endocrine surgery. Results are generally excellent, and morbidity and mortality are usually negligible. The operation requires proper identification of important structures such as the recurrent laryngeal nerve (RLN) and the parathyroid glands. Meticulous dissection and exhaustive hemostasis are important to ensure a dry field and to avoid inadvertent damage to the adjacent structures. The two most common techniques for hemostasis are suture ligatures and electrocoagulation. The use of electrocoagulation (EC) to control bleeding has the potential risk of injuring the surrounding structures from lateral dispersion of heat. New haemostatic techniques have been developed with the advent of laparoscopic surgery. Among other things, ultrasound instruments have been used for the dissection, division and coagulation of vessels and other tissue. Previous studies in Thyroidectomy observed a clinically and economically significant reduction in operating time with no increase in the complication rate when the Harmonic device has been used. The aim of the present clinical trial is to evaluate potential advantages of a new Harmonic device (FOCUS), developed especially for Thyroid procedures, in the use of HS in thyroidectomies when compared with EC in terms of operative time, number of ligatures, QoL, blood loss, pain intensity at the surgical site, amount of drainage, and complications, including the incidence of RLN palsy and hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Elected to undergo total thyroidectomy.
* Able to comprehend and sign the applicable study informed consent form.
* Able to return for all study mandated visits (visit 1 and 2)
* Be greater than or equal to 18 years of age.

Exclusion Criteria:

* Previous neck operation
* History of neck irritation
* Need for central or lateral compartment lymphadenectomy
* Patients under permanent pain killer medication
* Patients under anticoagulation medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive euthyroid patients with multinodular goiter for whom a total Thyroidectomy under general anesthesia is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Time incision to skin closure | during surgery

SECONDARY OUTCOMES:
Complications | intra- and postoperative

CONTACTS AND LOCATIONS:
Locations (2):
- CHU Sart-Tilman, Liège, Belgium
- University of Pisa, Pisa, Italy